CLINICAL TRIAL: NCT04274621
Title: The Application Value of Non-contact Infrared Thermometers in Temperature Screening in the General Population: a Real-world, Prospective, Observational Study
Brief Title: The Application Value of Non-contact Infrared Thermometers in Temperature Screening in the General Population
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WT2020-V1.0
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Non-contact Infrared Thermometer; Rapid Screening

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients, family members of patient, medical staff

SUMMARY:
The first epidemic of 2019 novel coronavirus (2019-nCoV)-infected pneumonia(NCIP) in Wuhan, China, has attracted global attention because of its strong transmission ability and certain fatality. Analyzing the clinical data of hospitalized patients with 2019-nCoV infection, the current studies found that fever, fatigue and dry cough were common symptoms, and 43.8% of the patients showed fever before admission. Some scholars emphasize that the most effective means to control the outbreak are early detection, early isolation, early diagnosis and early treatment. In the face of the pressure that a large number of people need rapid screening and the deficiency that the forehead temperature measurement is easily affected by the environment, the investigators would like to explore the accuracy and advantages of wrist temperature measurement in different environments and conditions in this period. And determine the thresholds of non-contact infrared thermometer for the screening of patients with fever, in order to provide clinical indicators for further detection of patients with suspected fever.

ELIGIBILITY:
Inclusion Criteria:

* patients, family members of patients, and medical staff

Exclusion Criteria:

* age <= 18 years
* Wearing hearing aid, having a cerumen
* Soft tissue infection, trauma patients
* Missing data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients, family members of patients, and medical staff
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
The Comparison of accuracy between wrist temperature and forehead temperature. | cross-sectional analyses in 2020
  The investigators used non-contact infrared thermometers to measure the value of wrist and forehead temperature in patients, family members of patients, medical staff. They record the value of temperature in the population and environment temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China